CLINICAL TRIAL: NCT06811454
Title: A Daily, Digital Mindfulness-Based Intervention for Depressive Symptoms After Serious Medical Illness
Brief Title: Mindfulness-based Intervention for Depressive Symptoms Sent Via Text (MINDSET)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CASE1Y24
Record Dates: First submitted 2025-01-31; First posted 2025-02-06 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Depression; Cancer; Stage III Breast Cancer; Stage II Breast Cancer; Stage I Breast Cancer; Stage III Prostate Cancer; Stage II Prostate Cancer; Stage I Prostate Cancer; Stage III Colorectal Cancer; Stage II Colorectal Cancer; Stage I Colorectal Cancer
Keywords: Post treatment Depression
MeSH Terms: conditions — Depression; Neoplasms; Breast Neoplasms; Prostatic Neoplasms; Colorectal Neoplasms | interventions — Stress Mindset Measure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ARM 1 (Experimental): Participants will be randomized to MINDSET
  Interventions: Behavioral: MINDSET
- ARM 2 (Other): Participants will be randomized to EUC
  Interventions: Behavioral: Enhanced Usual Care (EUC)

INTERVENTIONS:
Behavioral: MINDSET — Participants randomized to MINDSET will receive a text message at their preferred time each day for 8 weeks containing a link to the 15-minute audio content. At the end of each week (on day 7), participants will receive a second link to the weekly survey in the text. Participants will be able to play the audio content on their device by clicking the first link and access the weekly survey by clicking the second.
  Arms: ARM 1
Behavioral: Enhanced Usual Care (EUC) — Participants will receive a 1-page brochure summarizing publicly available information on depression self-care strategies via text each week for 8 weeks on the same day they receive the text message containing a link to the weekly survey (day 7). This information will come from the Facing Forward: Life After Cancer Treatment booklet from the National Cancer Institute.38 Weekly topics will include: 1) Reducing stress; 2) Coping with stress; 3) Coping with depression; 4) Feeling angry; 5) Feeling alone; 6) Finding meaning after treatment; 7) Social relationships; and 8) Seeking support. These materials do not include any content on mindfulness or cognitive therapy.
  Arms: ARM 2

SUMMARY:
The purpose of this study is to develop and test a new intervention to reduce depressive symptoms in post-treatment cancer participants.

DETAILED DESCRIPTION:
Mindfulness-based interventions (MBIs), including Mindfulness-based Cognitive Therapy (MBCT), reduce depressive symptoms in medically ill populations, including cancer survivors. However, MBIs have limitations, and if improved, could dramatically increase their clinical reach and impact. Most standardized MBIs are group-based, time intensive, difficult to scale, and can be costly. Thus, only a small portion of patients ever engage with MBIs. Digital approaches to delivering mindfulness content (apps and brief MBIs) have shown promise for addressing these barriers to accessibility and scalability. However, these digital approaches are not typically tailored for people with medical illness, like cancer, and/or have poor adherence. Mindfulness app user engagement decreases by 90% within 7 days of download, and the average total use of the app is only 16-21 minutes. Moreover, a recent review of MBIs that included standardized group-based MBIs (e.g., Mindfulness-Based Stress Reduction [MBSR]) and three mindfulness-based apps (e.g., Calm) estimated a 40-60% adherence rate of assigned at-home practice (30-45 minutes/day) in cancer survivors during the MBI, which further declines post-intervention. This suggests that the currently prescribed daily practice dosages are not feasible or accepted by this population. Thus, a brief MBI that optimizes the accessibility and scalability and other benefits of digital and asynchronous delivery, in a feasible and acceptable format, is critically needed for people with depressive symptoms and medical illness.

MBCT, adapted into a brief, daily and digitally delivered format, could increase access, scalability, acceptability, and adherence. While consistent practice for longer sessions yields the most benefit,21 studies have shown improved mood following 5 and 13 minutes of daily meditation for 2 and 8 weeks, respectively. Further, because creating and sustaining a new behavior, like daily meditation, requires consistent repetition, it is plausible that delivering content in short, digestible segments each day, as opposed to longer, weekly sessions, could improve adherence and sustain engagement. The full-length, 8-week MBCT protocol delivered digitally reduces depressive symptoms in cancer survivors, and the standardized 8-week MBCT protocol has already been abbreviated from 2- to 1-hour weekly groups (MBCT-Brief). When tested via remote delivery (telephone), MBCT-Brief showed a decrease in depressive symptoms in participants with medical illness (i.e., hypertension). Because of its abbreviated format and evidence for reducing depressive symptoms in people with medical illness, MBCT-Brief is a logical and feasible intervention to adapt into a daily text-delivered format for depressive symptoms in post-treatment cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

1. Self-reported mild to moderately-severe symptoms of depression (score 5-19 on PHQ-9).
2. A diagnosis of stage 0-III breast, prostate, or colorectal cancer.
3. Completion of primary cancer treatment within 2 years (excludes hormone therapy).
4. An ability to provide informed consent.
5. An ability to read and speak English.
6. Access to a web-enabled device (phone, tablet, computer).

Exclusion Criteria:

1. Self-reported minimal and severe depressive symptoms (<4 and > 20 on PHQ-9).
2. Self-reported suicidal ideation (>1 on item 9 PHQ-9).
3. Another psychological, medical, or other condition/issue determined that necessitates priority treatment and/or that would interfere with participation (e.g., schizophrenia, borderline personality disorder)
4. Current or recent substance abuse/dependence.
5. Stage IV cancer diagnosis.
6. A cancer recurrence actively requiring treatment.
7. Self-reported active mindfulness practice.
8. Prior participation in a formal mindfulness program (e.g., MBCT, Mindfulness-Based Stress Reduction Program, Mindfulness-Based Cancer Recovery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2026-08-03 (Estimated); Primary Completion 2028-03-31 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility as assessed by listening rate | 12 weeks
  80% listening rate of daily audio content
Feasibility as assessed by sample retention rate | 12 weeks
  80% sample retention
Acceptability rate as assessed by satisfaction rating of daily audio content | 12 weeks
  (>8 median satisfaction rating of daily audio content is measured as accepatble
Acceptability rate as assessed by Client Satisfaction Questionnaire (CSQ-8) post-MINDSET | 12 weeks
  >24 on the Client Satisfaction Questionnaire (CSQ-8) post-MINDSET will be considered as acceptable. CSQ-8 is a list of questions rating the satisfaction ranging from quite dissatisfied to very satisfied

SECONDARY OUTCOMES:
Symptoms of depression as measured by PROMIS-D-SF | 12 weeks
  The PROMIS-D-SF is an 8-question survey that measures depression on a scale from 1 (never) to 5 (always).
Symptoms of anxiety as measured by PROMIS-A-SF | 12 weeks
  The PROMIS-A-SF is an 8-question survey that measures anxiety on a scale from 1 (never) to 5 (always).

CONTACTS AND LOCATIONS:
Overall Officials: Chelsea Siwik, PhD, Principal Investigator — Case Comprehensive Cancer Center, Cleveland Clinic
Locations (1):
- Case Comprehensive Cancer Center, Cleveland Clinic Foundation, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
After the completion of the study and the associated publication, we will deposit de-identified data and metadata (i.e., codebook, focus group interview guides, protocols) that are necessary for or of sufficient quality to validate and replicate the research findings in the Open Science Framework repository (https://osf.io/).
Supporting Information: Study Protocol
Time Frame: Data will become available after the completion of the study and the associated publication and will remain available indefinitely.